CLINICAL TRIAL: NCT04621916
Title: A Multi-center, Prospective Study Evaluating the Rate of Inhibitor Recurrence Following Successful ITI in Patients Receiving Ongoing Once Per Weekly Factor VIII Therapy Along With Emicizumab and in Patients Who Discontinue FVIII Therapy and Are on Emicizumab for Prophylaxis
Brief Title: Preventing Inhibitor Recurrence Indefinitely
Acronym: PRIORITY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, Guy Young, MD, professor, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHLA-20-00189
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Hemophilia A; Immune Tolerance
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Emicizumab + FVIII weekly (Active Comparator): In addition to emicizumab prophylaxis,participants will receive non-prophylactic exposure to FVIII concentrates through weekly 50 IU/kg ±10% doses - the choice of FVIII concentrate is at the discretion of the PI.
  Interventions: Drug: FVIII; Drug: Emicizumab
- Emicizumab only (Active Comparator): Participants will only receive emicizumab prophylaxis.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: FVIII — This study will evaluate the inhibitor recurrence with or without ongoing FVIII exposure in patients with hemophilia A on emicizumab prophylaxis after a successful immune tolerance induction.
  Arms: Emicizumab + FVIII weekly
Drug: Emicizumab — This study will evaluate the inhibitor recurrence with or without ongoing FVIII exposure in patients with hemophilia A on emicizumab prophylaxis after a successful immune tolerance induction.

SUMMARY:
This study will enroll children who have hemophilia A with inhibitors who successfully completed immune tolerance induction per the ISTH criteria (negative inhibitor titer, recovery >66% of expected, and half-life of >6 hours with their current FVIII concentrate). Previous to emicizumab, there was only one option for these patients which was to continue FVIII therapy in a prophylaxis mode to prevent bleeding. There was a sense that the ongoing FVIII served to maintain tolerance however no evidence for this notion exists and in fact what limited data is available suggests that continuing FVIII may not be necessary simply to maintain tolerance.

To figure out this question, this will be a randomized, controlled 2 arm study which will randomize patients post-successful ITI to emicizumab plus weekly FVIII (for maintenance of tolerance) versus emicizumab alone. Patients will be followed for up to 2 years. We aim to enroll 52 subjects. The FVIII weekly arm can use any factor VIII concentrate and emicizumab is standard of care for inhibitor and non-inhibitor patients.

DETAILED DESCRIPTION:
Background & rationale: Hemophilia A is a serious life-long genetic bleeding disorder resulting from a mutation in the Factor VIII (FVIII) gene leading to abnormally low levels of FVIII. Treatment consists of replacing the missing FVIII with FVIII clotting factor concentrates (CFC). While FVIII CFC are very effective at preventing joint bleeding, they are immunogenic such that ~30% of patients develop anti-drug antibodies which neutralize the effect of the medications and are thus called inhibitors. Patients with inhibitors have worse morbidity and mortality as a result of increased and more difficult to treat bleeding episodes. Therefore, the major goal of therapy for patients who develop these antibodies is eradication of the inhibitor. The only approach that has been shown to be effective is called immune tolerance induction (ITI), and as its name implies, the purpose is to induce the patient's immune system to no longer make the inhibitors. Immune tolerance induction involves administering FVIII CFC on a regular and often intensive (daily) schedule for many months if not years. It can be effective, however, with successful ITI ranging from 40-90% in numerous previous studies. there exists a sizable minority of patients (~20-25% of all hemophilia A patients) who are ITI successes. For these patients, ongoing FVIII therapy has been the standard of treatment although once tolerization has been achieved, the treatment modality reverts to prophylaxis, however the continued regular exposure to prophylaxis is felt to also serve the purpose of maintaining tolerance.there is little to no data on whether ongoing FVIII exposure is required to maintain tolerance, and it is entirely possible that patients can discontinue routine factor therapy and not have a recurrence of their inhibitor. Only one study has even addressed this issue, and it found that inhibitor recurrence rates were the same among a group of tolerized patients who were subsequently adherent to a prophylaxis regimen and another group who were not adherent and therefore not receiving regular FVIII exposure.

While historically, this was a moot issue since the only appropriate therapy for severe hemophilia patients following successful ITI was to be prescribed FVIII prophylaxis, the recent licensure of a new medication has now made this question and knowledge gap very important. Emicizumab (Hemlibra, Roche, Basel, Switzerland) is a novel, bispecific, monoclonal antibody which can substitute for the function of activated FVIII by bringing activated factor IX and factor X into proper alignment and induce the formation of activated factor X.

Despite the high degree of efficacy of emicizumab for bleed prevention in inhibitor patients, the hemophilia community has still largely taken the stance that inhibitor eradication is a vital goal for any child who develops an inhibitor. The issue that the advent of emicizumab has raised, however, is what to do following successful ITI. As stated, traditionally, patients would continue FVIII therapy in the form of prophylaxis and the question of loss of tolerance and inhibitor recurrence was moot, however given the advantages of emicizumab, it is likely that many patients/parents will not accept continuing with the need for repeated intravenous infusions (and central venous catheters in many children) when an alternative agent with excellent efficacy and a much lower treatment burden exists. Thus, objective of this study is to determine whether ongoing factor VIII therapy is required for maintenance of tolerance.

Study population: patients who have undergone successful ITI and are currently on emicizumab or willing to be on emicizumab.

Study methodology: This will be a prospective, randomized trial of weekly FVIII CFC therapy versus no routine FVIII therapy for patients who have undergone successful ITI and are currently on emicizumab or willing to be on emicizumab.

Description of study arms: Group 1 will receive ongoing once per weekly factor VIII therapy along with emicizumab after completion of a successful ITI. Group 2 will discontinue FVIII therapy and are on emicizumab for prophylaxis after completion of a successful ITI.

Study endpoints: Study endpoints are to find out the number of subjects that maintained immune tolerance with/without FVIII exposure, understand the need for FVIII exposure for maintaining immune tolerance and to estimate the treatment burden and the cost effectivity for ongoing FVIII exposure after a successful ITI.

Follow-up: Patients will be seen every month for inhibitor recurrence until 4th month of the study, and every two months until the first year of the study, at 18th month and at the end of the study. If there is a bleeding episode or an inhibitor, then there will be an unscheduled visit.

Statistics: Patients will be categorized as either having a recurrence of an inhibitor or not. Thus, a 2x2 Chi-square contingency table will be able to group the subjects into those who received ongoing factor VIII and those who did not and those who did versus those who did not have an inhibitor recurrence. Fisher's exact test will be used to calculate the difference in proportion between the groups (inhibitor-positive and inhibitor-negative).

Plans for analysis: Our goal is to complete the project including a submission for an abstract and publication within 24 months from the start of patient accrual.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤12 years at the time of signing the informed consent
* Male patients with severe (<1%) or moderate (<2%) hemophilia A
* History of a high titer (>5 BU) inhibitor
* Within 1 year of successful ITI, according to ISTH definitions (inhibitor titer <0.6 BU, recovery more than 60% of expected, and half-life of >6 hours). Successful ITI has been achieved with any FVIII concentrate.
* Currently on emicizumab or willing to alter their prophylaxis treatment to emicizumab per study protocol.

Exclusion Criteria:

* Age >12 years at the time of signing the informed consent
* Partial tolerance (not meeting criteria for complete tolerance per ISTH)
* History of anti-drug antibodies to emicizumab
* Unwilling to receive exposure to intravenous FVIII concentrates.
* History per the investigator's discretion of non-compliance to prior therapy.

Ages: 0 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Since Hemophilia is a X-linked bleeding disorder occurring mostly in males we expected to mostly enroll male-identified subjects.
Enrollment: 52 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Inhibitor recurrence | The goal is to complete all study procedures in 2 years.
  FVIII inhibitor level will be checked on certain time points during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Young, MD, Principal Investigator — Professor of Pediatrics, Director of Hemostasis and Thrombosis Center
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be in the results of the study publication.
Supporting Information: Study Protocol